CLINICAL TRIAL: NCT06487767
Title: The Validity of the Use of Imaging in Cervical Cancer Staging
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pretoria (Other)
Collaborators: Dr Edwin Mnisi (Unknown); Prof Mike Sathekge (Unknown); Prof N Khan (Unknown)
Responsible Party: Principal Investigator, Leon Snyman, Professor, University of Pretoria
Other Study IDs: 704/2023
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer Stage, Imaging Modalities
Keywords: Cervical cancer; Ultrasound; MRI; CT Scan; PET-CT scan
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surgery — Surgery for operable cervical cancer

SUMMARY:
The study wil aim to investigate the accuracy of imaging in the staging of women diagnosed with cervical cancer

DETAILED DESCRIPTION:
Patients with cervical cancer undergoing surgery will also undergo PET-CT scan, CT scan, trans-abdominal ultrasound of the pelvis and abdomen to assess pelvic and para-aortic lymph node status, MRI and trans-vaginal ultrasound (TVUS) to assess tumour size and parametrial infiltration. As per the current unit protocol, patients will be assessed clinically for operability. The performance of the different imaging modalities will be measured against the histological status of the parametric and lymph nodes and tumour size as measured by the pathologists.

CT, PET-CT, MRI and abdominal ultrasound will be reported as per the usual departmental process. Staff in the radiology department will be blinded for the different imaging modalities performed. TVUS will be performed in the unit by different gynaecological oncologists and fellows and at the time of the investigation will be blinded with regards to clinical findings and the reports of other imaging studies performed.

The sensitivity, specificity, positive and negative predictive values will be calculated for the different imaging modalities.

ELIGIBILITY:
Inclusion Criteria:

- Women diagnosed with cervical cancer Able and willing to provide informed consent

Exclusion Criteria:

Previously treated for cervical cancer Unable to provide informed consent Patients with contra-indications to undergo surgical treatment

-

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women diagnosed with cervical cancer
Study Population: Women diagnosed with cervical cancer scheduled for surgical treatment or intervention
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | 2 years
  Metrics of imaging

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Visser, MSc, Study Director — Trial administrator
Locations (1):
- Kalafong Provincial Tertiary Hospital, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No